CLINICAL TRIAL: NCT02053961
Title: The Efficacy of dTMS Among Patient Who Suffer From Tinnitus
Brief Title: Deep TMS of the Left Auditory Cortex Using the HMCIPCC Coil, in the Treatment of Patients With Tinnitus.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: dTMS-Tinnitus- wolfson
Record Dates: First submitted 2014-01-28; First posted 2014-02-04 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1Hz dTMS Real (Active Comparator): This group will receive dTMS real treatment of 1Hz
  Interventions: Device: Deep Transcranial Magnetic Stimulation
- 1HZ dTMS SHAM (Sham Comparator): This group will receive 1HZ dTMS SHAM treatment
  Interventions: Device: Deep Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Deep Transcranial Magnetic Stimulation — 1Hz dTMS real treatment
Device: Deep Transcranial Magnetic Stimulation — 1Hz dTMS SHAM treatment
  Arms: 1HZ dTMS SHAM

SUMMARY:
The study is a double-blind study designed to evaluate the efficacy of deep transcranial magnetic stimulation (deep TMS) of the left auditory cortex using the HMCIPCC coil, in the treatment of patients with tinnitus

DETAILED DESCRIPTION:
Stages of the study:

A. Patient recruitment stage: hearing tests battery including: otoscopy, tympanometry, pure-tone audiometry - 0 to 20 dB HL; 21 to 60 dB HL and more than 60 dB HL, tinnitus matching, TQ and VAS.

B. Patients will be assign to one of two study groups, Deep TMS over the left auditory cortex and Sham. .

C. TMS Acute treatment phase:

TMS treatment will be administer for two weeks: 5 days a week for half an hour. Before each TMS treatment session, patients will undergo training exercises designed to stimulate the neural network associated with attention processes Monitoring for evaluation of treatment efficacy and side effects will be perform on a daily basis. . The overall time of each session is estimate to be 1 hour.

D. TMS Maintenance phase:

Four additional TMS treatment sessions will be administered once weekly for another 4 weeks.

Long-term durability of treatment effect will be assessed up to 90 days after the last TMS session.

E. TMS treatment program:

1. The subject will be required to use earplugs to minimize risk of hearing impairment.
2. Motor threshold stimulation intensity will be determined prior to each TMS session. .
3. Subjects will receive either active TMS or sham treatment, depending on the experimental group to which they were assign. During the first 2 weeks, five treatment sessions will be administer each week. During the following 4 weeks, one treatment will be administer weekly. Overall, each subject will receive 16 TMS session in 6 treatment weeks.

F. Safety:

Throughout the trial subjects will be constantly monitored by a physician. Any adverse effect or subjective discomfort experienced will be documented and addressed.

Magnetic stimulation treatment will be administered by an operator trained and certified by Brainsway.

Subjects who wish to withdraw from the study will be free to do so at any point.

Drugs belonging to benzodiazepine class will be permitted if necessary at daily doses up to the equivalent of 2 mg Lorazepam (Lorivan).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 20-70.
2. Self-report of tinnitus in one or both ears, persisting for over a year, with no other hearing impairment.
3. Mild/moderate/severe tinnitus. Severity of tinnitus will be diagnosed using the TQ (Goebel & Hiller) / the THI (Newman & Jacobson).
4. Unresponsive to standard tinnitus medication.
5. Normal results on pure tone audiometry testing (threshold ≤ 25 dB hearing level in all frequencies from 250 to 8000 Hz).
6. Normal middle ear status was demonstrated by tympanometry, stapedius reflex tests, and otoscopy.
7. Normal results on neurological and physiological examinations.
8. Gave their oral and written consent to participate in the trial.

Exclusion Criteria:

1. A DSM-IV Axis-I psychiatric disorder.
2. Use of medication that may be a risk factor for seizures, such as:

   antipsychotic medication; high dosage of antidepressant medication; drugs belonging to benzodiazepine class will be permitted if necessary at daily doses up to the equivalent of 2 mg Lorazepam (Lorivan)' any other drug that is considered a risk factor for seizures by the Principal Investigator.
3. History of intolerance to TMS.
4. Diagnosis of a severe personality disorder according to the DSM-IV.
5. Current suicidal ideation.
6. Uncontrolled hypertension.
7. History of epilepsy, seizure, or heat convulsion.
8. History of epilepsy or seizure in first degree relatives.
9. History of head injury or stroke.
10. History of any metallic particles in the head (except dental fillings).
11. History of surgery entailing metallic implants or known history of any metallic particles in the eye, implanted cardiac pacemakers, cochlear implants, use of neurostimulators, or any medical pumps.
12. History of drug or alcohol abuse.
13. Inability to communicate adequately with examiner.
14. Participation in another clinical study, either concurrent with this trial or in the 3 months preceding it.
15. Inability to sign a consent form.
16. Pregnancy or inadequate birth control.
17. Severe hearing impairment.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01 (Estimated); Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
TQ - Tinnitus questionnaire | 90 days after the last treatment session

SECONDARY OUTCOMES:
VAS (100 - worst possible tinnitus related discomfort; 0 - wellness) | baseline, week 1: day 1-5, and week 2: day 1-5

CONTACTS AND LOCATIONS:
Overall Officials: Yair Lampel, Prof., Principal Investigator — Neurology Department, Wolfson Hospital, Israel
Locations (1):
- Wolfson Hospital, Holon, Israel